CLINICAL TRIAL: NCT00525629
Title: The Metabolic Effects of Short-term Walnut Consumption in Subjects With the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christos Mantzoros (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor-Investigator, Christos Mantzoros, Principal Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2006P000255
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-06

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnut Diet (Experimental): 48 Grams of Walnuts Daily
  Interventions: Dietary Supplement: Walnuts
- Control Diet (Placebo Comparator): Isocaloric Diet with No Walnuts
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Walnuts — 48 Grams of Walnuts Daily
  Arms: Walnut Diet
Dietary Supplement: Control — Control Diet with No Walnuts
  Arms: Control Diet

SUMMARY:
Walnuts include many potentially beneficial micronutrients and phytochemicals, in this study we propose to examine the effects of walnuts independent of macronutrient content. The purpose of this proposal is to study in depth the short-term effects of walnut consumption in men and women with the metabolic syndrome.

Study Aim 1: To investigate the effects of walnuts (48gms per day over 3 days) on insulin resistance in subjects with the metabolic syndrome.

Study Aim 2: To investigate the effects of 48gms per day of walnuts over 3 days on lipids and inflammatory markers.

Study Aim 3: To assess the possible mechanisms of the biological effects of short-term walnut consumption through assessment of adipokines, resting metabolic rate, gene expression in white blood cells and the effect of walnuts when consumed as part of a mixed meal, on glucose excursions, insulin secretion and the excretion of gut peptides and free fatty acids.

DETAILED DESCRIPTION:
During the whole study period, you will be asked to maintain a constant body weight and you will receive advice from the dietitian regarding a weight stable diet and exercise pattern. You will also be asked to avoid walnuts during the entire study period. The intervention and the measurements during each of the visits are described below.

If you agree to be in this study, you will be asked to read and sign this consent form. After you sign the consent form, the following things will happen:

1. Screening Procedures: Screening procedures are tests and procedures that will be done to determine if you are eligible to take part in the research study. For this research study, the screening procedures include:

   1. A detailed medical history and interview about lifestyle factors and medication use
   2. A brief physical examination to document any abnormalities in your body appearance and measurement of weight, height and waist circumference.
   3. Drawing of blood from the forearm for fasting blood glucose (blood sugar), lipid profile (cholesterol and other fats in blood), creatinine (a measure of your kidney function), and complete blood count (CBC).
   4. Collection of urine for a HCG pregnancy test (women only)

   For the blood tests, you will be asked not to eat or drink anything (except water) from 8 pm the previous evening until you arrive for the study visit the following morning.

   Samples of your blood will be stored under code to be used for future research by the BIDMC investigators but your name will not be identified. If for any reason you have decided to withdraw from the study or if you have not met the criteria for enrollment into the study, all the blood drawn at the screening visit will be discarded.

   Next, you will meet with a research dietician to receive instructions for the 2-week run-in period (see below).
2. Randomization Procedures:

   You will be randomly assigned (like the flip of a coin) to receive either walnut containing milkshake or placebo containing milkshake on your first visit. Each participant will receive walnut containing milkshake during one visit and a milkshake that looks and tastes the same but without walnuts (placebo) on the other visit but the order of the visits will be randomized.
3. Research Procedures: If you qualify to take part in this research study, you will undergo these research procedures:

   Run-in period:

   You will meet with a research dietician who will provide instructions about maintaining your normal diet and physical activity pattern and about avoiding walnut-containing foods and drinks.

   Study Visit 1 and 2 Each study visit involves a 4-day (4 overnight) stay at the General Clinical Research Center. You will be admitted at 9pm the evening before the first day of the visit. You will be asked to complete a hunger questionnaire each morning before you have had anything to eat. You will receive a milkshake each morning containing either with or without walnuts. We will repeat the hunger questionnaire before your lunch each day. You will be provided with lunch and dinner based on what you like to eat. The calorie content of the lunch and dinner will be controlled so that you will neither gain or lose weight during your stay.

   Day 1 The following morning the following tests will be performed; Measure your weight, waist circumference, and blood pressure. Resting Metabolic Rate Fasting blood tests Body composition Mixed meal challenge You will receive your first milkshake as part of the mixed meal challenge.

   Day 2 On day 2 there is no testing but you will complete the hunger questionnaire and receive another milkshake for breakfast.

   Day 3

   On day 3 you will have the following tests performed:

   Insulin Suppression Test Fasting blood sample At the end of the insulin suppression test, you will receive another milkshake.

   Day 4 On the morning of your last day you will have repeat testing as on the first day of the visit and will leave the hospital at mid-day after the testing is complete.

   Washout phase Between the 2 study visits you will enter a washout phase where you will continue your normal healthy diet and exercise but avoid walnuts in your diet. After 1 month of washout you will return to the GCRC for your second study visit.
4. Tests performed during the study

Resting Metabolic Rate RMR is the amount of calories you burn without doing any physical work. Your RMR will be measured with a commonly used instrument. You will be asked to lie quietly in bed and stay awake with a large plastic hood over your head and upper body for about 20 minutes and breathe normally while the air you breathe out is being collected.

Fasting blood tests Blood samples will be used to measure sugar, insulin levels, lipids (LDL, HDL, and total cholesterol, triglycerides), hormones (such as leptin, resistin and adiponectin) and blood markers of inflammation (such as TNF and CRP). We will also perform a blood test to measure the expression of genes involved in metabolism in your white blood cells. For the blood tests, you will be asked not to eat or drink anything (except water) from 8 pm the previous evening until. In addition, you will be asked not to participate in vigorous physical activity on the day before the visit. Samples of your blood will be stored under code to be used for future related blood measurements by the BIDMC investigators but your name will not be identified.

Body composition To measure the amount of fat in your body we will use bioelectrical impedance analysis. During this procedure you will lie down and the speed of an electric signal through your body will be measured. This signal is not painful.

Mixed meal challenge You will have a small catheter (a small plastic tube) placed in a vein with a needle in your forearm to draw blood. This will prevent the need for multiple needle sticks for the required blood draws. The catheter will be taped to stay in place for approximately three hours. You will drink a milkshake and your blood will be drawn through the catheter 15 min after the milkshake is given and then at 30-minute intervals for 3 hours to measure how you metabolize the nutrient drink.

Insulin Suppression Test (also called Galvin's Index) This test consists of an overnight fast (nothing to eat or drink after 11pm the night before), after which two IV lines will be placed in your arms. Glucose, insulin,octreotide (a hormone commonly used in clinical practice for treating several different diseases) and albumin ( a protein found in blood) will be infused through the IV. Blood samples will be drawn through the other IV line at times -10 minutes, 0 minutes, and every 30 minutes for two and a half hours, then every 10 minutes for an additional 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome is defined as follows:

Central Obesity- for Europid men this is a waist circumference of > 94cm for women >80cm or BMI >30.

Plus 2 of the following 4 factors

1. Elevated triglycerides: > 150 mg/dL
2. Reduced HDL cholesterol < 40 mg/dL in men and < 50 mg/dL in women.
3. Raised diastolic blood pressure systolic BP > 130mmHg or diastolic BP > 85mmHg or treatment with antihypertensives.
4. Raised fasting plasma glucose > 100mg/dL or previously diagnosed type II diabetes.

Exclusion Criteria:

1. Subjects with diabetes requiring medication or insulin are excluded.
2. Subjects with any medical condition or on any treatment, which would interfere with the study outcomes or would make participation potentially harmful such as pregnancy or breastfeeding, anemia, heart disease, stroke, malabsorption syndromes according to a detailed medical history.
3. Present alcoholism or drug abuse or use of medications that could interfere with the study such as corticosteroids, growth hormone, antiretroviral therapy. These conditions will be screened for by a detailed history and systems review.
4. Individuals with nut allergy are excluded.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brennan AM, Sweeney LL, Liu X, Mantzoros CS. Walnut consumption increases satiation but has no effect on insulin resistance or the metabolic profile over a 4-day period. Obesity (Silver Spring). 2010 Jun;18(6):1176-82. doi: 10.1038/oby.2009.409. Epub 2009 Nov 12. PMID 19910942

RESULTS

PARTICIPANT FLOW:
Groups:
- Walnut Diet First, Then Control Diet: patients were asked to consume 48g of walnuts per day
- Control Diet First, Then Walnut di: patients were asked to consume an isocaloric Diet with no Nuts
Period: First Intervention
Arm/Group | Walnut Diet First, Then Control Diet | Control Diet First, Then Walnut di
Started | 20 | 20
Completed | 15 | 15
Not Completed | 5 | 5
Period: Washout
Arm/Group | Walnut Diet First, Then Control Diet | Control Diet First, Then Walnut di
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Walnut Diet First, Then Control Diet | Control Diet First, Then Walnut di
Started | 15 | 15
Completed | 0 | 0
Not Completed | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients received both interventions and are included in this group analysis
Arm/Group | All Patients
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 37.1 (1.4)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 207 (11.8)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 199.2 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance
Description: HOMA-IR (homeostatic model assessment of insulin resistance) given in units as it is a ratio equation.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: HOMA-IR index
Arm/Group | Walnut Diet | Control Diet
Number analyzed (Participants) | 30 | 30
HOMA-IR index | 6.06 (3.78) | 5.72 (2.7)

ADVERSE EVENTS:
Time Frame: 4 days (during the study)
Description: Adverse events were reported in real time, as they occurred (if any) by a physician who saw the patients each day. As this was a dietary analysis/no pharmacological intervention, no adverse events were expected.
Groups:
- Walnut Diet: 48g of walnuts per day
- Control Diet: Isocaloric Diet with no Nuts.
Arm/Group | Walnut Diet | Control Diet
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No